CLINICAL TRIAL: NCT06915727
Title: Pafolacianine for Localization of Pediatric Extracranial Solid Tumors
Brief Title: An Imaging Agent (Pafolacianine) for Identifying Lesions in Pediatric Patients With Primary or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC250701; NCI-2025-02149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-012249 (Other: Mayo Clinic Institutional Review Board); MC250701 (Other: Mayo Clinic)
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Childhood Malignant Solid Neoplasm; Childhood Malignant Thoracic Neoplasm; Malignant Abdominal Neoplasm; Malignant Neck Neoplasm; Malignant Pelvic Neoplasm; Metastatic Childhood Malignant Solid Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms; Pelvic Neoplasms | interventions — Specimen Handling; Pafolacianine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (pafolacianine + NIR) (Experimental): Patients receive pafolacianine IV over 60 to 90 minutes and undergo NIR fluorescent imaging during standard of care (SOC) surgery on study. Patients also undergo collection of tissue during SOC surgery on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Near Infrared Imaging; Drug: Pafolacianine Sodium; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Near Infrared Imaging — Undergo NIR fluorescent imaging
  Other Names: Near-Infrared Imaging; NIR Imaging
Drug: Pafolacianine Sodium — Given IV
  Other Names: Cytalux
Procedure: Surgical Procedure — Undergo SOC surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, Not Otherwise Specified (NOS); Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery; Surgery, NOS

SUMMARY:
This phase III trial studies how well pafolacianine works for identifying cancerous lesions in children and adolescent patients with primary solid tumors or solid tumors that have spread from where they first started (primary site) to other places in the body (metastatic). Pafolacianine is a fluorescent imaging agent that targets folate receptors which are overexpressed in many cancers and is used with near infrared (NIR) imaging during surgery to identify tumor cells. NIR uses a special camera that uses wavelengths in the infrared range to visualize and locate the tumor cells that are lit up by the pafolacianine. Giving pafolacianine for NIR imaging may work better than other imaging agents in identifying cancerous lesions in pediatric patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Willingness of research participant or legal guardian/representative to give written informed consent
* Age 6 months to 17 years
* Have a diagnosis, or a high clinical suspicion, of a solid tumor in the neck, chest, abdomen, pelvis, or extremities with a plan for surgical resection including embryonal tumors, sarcomas, neurogenic tumors, carcinomas, mesenchymal tumors, germ cell tumors. Children may undergo surgical resection or biopsy of a solid tumor that is suspected to be malignant without a separate preoperative biopsy; therefore, the tumor type may not be definitively known preoperatively

Exclusion Criteria:

* Previous exposure to Cytalux™ (pafolacianine) injection
* Any medical condition that in the judgement of the investigators could potentially jeopardize the safety of the participant
* History of anaphylactic reactions to products containing indocyanine green for near infrared imaging. Participants with a medical history of 'idiopathic anaphylaxis' will require evaluation
* History of allergy to any of the components of Cytalux™ (pafolacianine) injection
* Presence of any psychological, familial, sociological condition or geographical challenges potentially hampering compliance with the study protocol or follow-up schedule
* Received an investigational agent in another investigational drug or vaccine trial within 30 days prior to the administration of the study drug. Investigational trials involving administration of drugs or vaccines which are already Food and Drug Administration (FDA)-approved, such as Children's Oncology Group cooperative trials, are okay
* Known sensitivity to fluorescent light
* Pregnancy
* Unable or unwilling to discontinue folic acid, folate supplements, and multi-vitamins containing folate 48 hours prior to drug administration
* Renal failure on dialysis or estimated glomerular filtration rate (eGFR) < 30 mL/min/1.72m^2 as measured by the U25 eGFR equation for patients ≥1 year(s) of age. For patients < 1 year of age, creatinine > 2x the upper limit of normal will serve as an exclusion criteria. Creatinine will be measured by enzymatic assay with calibration traceable to the international standard reference materials and minimal bias compared to isotope-dilution mass spectrometry (IDMS) reference methodology.
* Undergoing workup for liver failure or listed for liver transplant. Patients with Gilbert's syndrome will be excluded if impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin
* Unable or unwilling to use adequate birth control/contraceptive measures or abstain from sexual activity for 30 days following the study intervention
* Anticipated need to donate ova or sperm within 30 days following study intervention

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Cytalux™ (pafolacianine) injection used with NIR fluorescent imaging for detecting lesions | Up to 30 days after surgery
  Each excised specimen will be analyzed for histologic findings to determine accuracy of Cytalux™ (pafolacianine) injection used with near infrared (NIR) fluorescent imaging for detecting lesions. Accuracy will be assessed using sensitivity and specificity.

SECONDARY OUTCOMES:
Time between Cytalux™ administration and NIR imaging detection intraoperatively | Day 0 to 1
  Descriptive statistics will be performed and descriptive summaries such as mean (standard deviation) or median (minimum, maximum) for continuous variables and frequencies and percentages for categorical variables will be reported.
Reasons for not excising NIR avid lesions | Day 0 to 1
  Descriptive statistics will be performed and descriptive summaries such as mean (standard deviation) or median (minimum, maximum) for continuous variables and frequencies and percentages for categorical variables will be reported. All tests will be two sided and p-values less than 0.05 will be considered statistically significant.
Incidence of Adverse Events surgery | From study enrollment up to 30 days after surgery
  Cytalux™ (pafolacianine) will be assessed for safety in children and adolescent patients undergoing by the number and severity of adverse events (AEs), defined as events (serious or non-serious) of scientific and medical concern specific to the investigational product and/or the combination of products being used in a study. AEs will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie F. Polites, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials